CLINICAL TRIAL: NCT06173297
Title: Assessing the Agreement Between Endoscopic and Histopathological Diagnosis of Colorectal Sessile Serrated Lesions.
Status: Completed | Type: Observational
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Sponsor
Other Study IDs: AVAP-NG 1415
Record Dates: First submitted 2023-12-04; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Sessile Serrated Adenoma; Colorectal Polyp; Adenoma Colon; Colorectal Cancer; Colonoscopy; Adenoma Detection Rate; Quality Indicator
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study was to assess the degree of agreement between the endoscopic and anatomopathological diagnosis of sessile serrated colorectal lesions in adult patients undergoing colonoscopy in Hospital Sírio-Libanes.

The main questions it aimed to answer were:

* The degree of agreement between endoscopic and anatomopathological diagnosis of sessile serrated colorectal lesions by calculating the Kappa Value of agreement.
* To establish the detection rate of sessile serrated lesions and adenomas in the Endoscopy Department at Hospital Sírio-Libanês.
* To evaluate the degree of agreement between endoscopic and anatomopathological diagnosis of sessile serrated colorectal lesions based on the resection method.
* To assess the accuracy, positive predictive value, and negative predictive value of endoscopic diagnosis of serrated lesions compared to anatomopathological diagnosis.

The data were prospectively collected through a form specifically designed for this project, that was completed immediately after the examination by the performing colonoscopist. All patients enrolled in this study agreed to participate in it and signed an informed consent form prior to the colonoscopy.

DETAILED DESCRIPTION:
The study population was:

Patients aged over 18 undergoing colonoscopy at Hospital Sírio-Libanês in the Bela-Vista unit, São Paulo, Brazil, between June and August 2020.

The sample:

For the present study, an odds ratio of 1.5 in the adenoma detection rate of colorectal lesions was considered concerning the vascular pattern classification of the lesion (NICE), with an expected discordance rate of 30% regarding the histopathological pattern. To achieve this, an estimated sample size of 758 patients was calculated, considering an 80% statistical power and a risk α≤5% for a Type I error, using the McNemar's test for proportions.

Inclusion criteria:

* Patients undergoing elective colonoscopy at Hospital Sírio-Libanês between February 2020 and August 2020.
* Age over 18 years.

Exclusion criteria:

* Patients with inflammatory bowel disease (IBD)
* Patients diagnosed with hereditary polyposis or non-polyposis syndromes.
* Patients with a history of colorectal surgery.
* Patients previously diagnosed with colorectal cancer (CRC).

Study variables analyzed:

* Age (years)
* Gender
* Colon preparation (Boston Scale)
* Presence of colorectal lesions
* Lesion resection technique
* Lesion size
* Lesion location
* Morphological classification of the lesion (Paris)
* Vascular pattern classification of the lesion (NICE)
* Number of lesions found per examination/patient.

Methods:

All colonoscopies in this study were conducted in the endoscopy department of Hospital Sírio-Libanês, and the equipment used was the Olympus™ EVIS Exera III - CV190.

All lesions identified in the study were sent to the pathology service of Hospital Sírio-Libanês for specialized and standardized anatomopathological analysis. The pathologists were blinded to the endoscopic diagnosis of the lesions. The lesions were classified according to the 2019 WHO Classification and subsequently categorized for this study into: hyperplastic polyps, adenomas, sessile serrated lesions, adenocarcinoma, or "others".

Statistical analysis:

Data obtained was assessed using the Gaussian curve and determined as parametric or non-parametric using the Kolmogorov-Smirnov test and the Shapiro-Wilk test. Parametric data were represented by mean and standard deviation, while non-parametric data were represented by median and interquartile range (25th and 75th percentiles). Categorical data were represented by absolute frequency (n) and relative frequency (%) and presented through contingency tables.

Sensitivity, specificity, positive predictive values, and negative predictive values (with corresponding 95% confidence intervals) of colonoscopy for diagnosing sessile serrated lesions using the anatomopathological examination as the gold standard were calculated.

To evaluate agreement between colonoscopy diagnosis and anatomopathological diagnosis, both overall and according to the resection method employed, Cohen's Kappa coefficients and their respective 95% confidence intervals were calculated. These coefficients were then categorized based on Landis & Koch's criteria (1977).

Ethical considerations:

The research project for this study was thoroughly detailed and submitted for analysis to the Research Ethics Committee (CEP) of Hospital Sírio-Libanês, receiving approval under CAAE 27604919.2.0000.5461. Patients participating in the study agreed to take part and signed the Informed Consent Form. The involved colonoscopists committed to maintaining the confidentiality of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colonoscopy at Hospital Sírio-Libanês between February 2020 and August 2020.
* Age over 18 years.

Exclusion Criteria:

* Patients with inflammatory bowel disease (IBD)
* Patients diagnosed with hereditary polyposis or non-polyposis syndromes.
* Patients with a history of colorectal surgery.
* Patients previously diagnosed with colorectal cancer (CRC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 undergoing colonoscopy at Hospital Sírio-Libanês in the Bela-Vista unit, São Paulo, Brazil, between June and August of 2020.
Sampling Method: Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
To assess the degree of agreement between the endoscopic and the anatomopathological diagnosis of sessile serrated colorectal lesions | 2 years
  To evaluate concordance between colonoscopy diagnosis and anatomopathological diagnosis, both overall and according to the resection method employed, Cohen's Kappa coefficients and their respective 95% confidence intervals were calculated. These coefficients were then categorized based on Landis & Koch's criteria (1977).

SECONDARY OUTCOMES:
To establish the detection rate of sessile serrated lesions and adenomas in the Endoscopy Department at Hospital Sírio-Libanês. | 2 years
  The Detection Rate in colonoscopy is calculated by dividing the number of procedures where at least one of the interested lesion is detected by the total number of procedures performed by the colonoscopist, and then multiplying by 100 to get a percentage.
Evaluate the degree of agreement between endoscopic and anatomopathological diagnosis of sessile serrated colorectal lesions based on the resection method. | 2 years
  To evaluate concordance between colonoscopy diagnosis and anatomopathological diagnosis, both overall and according to the resection method employed, Cohen's Kappa coefficients and their respective 95% confidence intervals were calculated. These coefficients were then categorized based on Landis & Koch's criteria (1977).
Assess the accuracy, positive predictive value, and negative predictive value of endoscopic diagnosis of serrated lesions compared to anatomopathological diagnosis. | 2 years
  Sensitivity, specificity, positive predictive values, and negative predictive values (with corresponding 95% confidence intervals) of colonoscopy for diagnosing sessile serrated lesions using the anatomopathological examination as the gold standard were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela S Oliveira, Master, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sírio-Libanes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Pan J, Xin L, Ma YF, Hu LH, Li ZS. Colonoscopy Reduces Colorectal Cancer Incidence and Mortality in Patients With Non-Malignant Findings: A Meta-Analysis. Am J Gastroenterol. 2016 Mar;111(3):355-65. doi: 10.1038/ajg.2015.418. Epub 2016 Jan 12. PMID 26753884
- [Background] Kaminski MF, Robertson DJ, Senore C, Rex DK. Optimizing the Quality of Colorectal Cancer Screening Worldwide. Gastroenterology. 2020 Jan;158(2):404-417. doi: 10.1053/j.gastro.2019.11.026. Epub 2019 Nov 20. PMID 31759062
- [Background] Wolf AMD, Fontham ETH, Church TR, Flowers CR, Guerra CE, LaMonte SJ, Etzioni R, McKenna MT, Oeffinger KC, Shih YT, Walter LC, Andrews KS, Brawley OW, Brooks D, Fedewa SA, Manassaram-Baptiste D, Siegel RL, Wender RC, Smith RA. Colorectal cancer screening for average-risk adults: 2018 guideline update from the American Cancer Society. CA Cancer J Clin. 2018 Jul;68(4):250-281. doi: 10.3322/caac.21457. Epub 2018 May 30. PMID 29846947
- [Background] Brenner H, Hoffmeister M, Arndt V, Stegmaier C, Altenhofen L, Haug U. Protection from right- and left-sided colorectal neoplasms after colonoscopy: population-based study. J Natl Cancer Inst. 2010 Jan 20;102(2):89-95. doi: 10.1093/jnci/djp436. Epub 2009 Dec 30. PMID 20042716
- [Background] Hassan C, Antonelli G, Dumonceau JM, Regula J, Bretthauer M, Chaussade S, Dekker E, Ferlitsch M, Gimeno-Garcia A, Jover R, Kalager M, Pellise M, Pox C, Ricciardiello L, Rutter M, Helsingen LM, Bleijenberg A, Senore C, van Hooft JE, Dinis-Ribeiro M, Quintero E. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 Aug;52(8):687-700. doi: 10.1055/a-1185-3109. Epub 2020 Jun 22. PMID 32572858
- [Background] O'Brien MJ, Winawer SJ, Zauber AG, Gottlieb LS, Sternberg SS, Diaz B, Dickersin GR, Ewing S, Geller S, Kasimian D, et al. The National Polyp Study. Patient and polyp characteristics associated with high-grade dysplasia in colorectal adenomas. Gastroenterology. 1990 Feb;98(2):371-9. PMID 2403953
- [Background] Mareth K, Gurm H, Madhoun MF. Endoscopic Recognition and Classification of Colorectal Polyps. Gastrointest Endosc Clin N Am. 2022 Apr;32(2):227-240. doi: 10.1016/j.giec.2021.12.003. Epub 2022 Feb 22. PMID 35361333
- [Background] Kim JH, Kang GH. Evolving pathologic concepts of serrated lesions of the colorectum. J Pathol Transl Med. 2020 Jul;54(4):276-289. doi: 10.4132/jptm.2020.04.15. Epub 2020 Jun 26. PMID 32580537
- [Background] Vennelaganti S, Cuatrecasas M, Vennalaganti P, Kennedy KF, Srinivasan S, Patil DT, Plesec T, Lanas A, Horndler C, Andraws N, Cherian R, Mathur S, Hassan C, Repici A, Klotz D, Musulen E, Risio M, Castells A, Gupta N, Sharma P. Interobserver Agreement Among Pathologists in the Differentiation of Sessile Serrated From Hyperplastic Polyps. Gastroenterology. 2021 Jan;160(1):452-454.e1. doi: 10.1053/j.gastro.2020.09.015. Epub 2020 Sep 18. No abstract available. PMID 32950521
- [Result] Ahmad A, Moorghen M, Wilson A, Saunders BP. NBI International Colorectal Endoscopic-derived high-confidence optical diagnosis of small polyps compared with histology: understanding errors to improve diagnostic accuracy. Gastrointest Endosc. 2023 Jan;97(1):78-88. doi: 10.1016/j.gie.2022.08.032. Epub 2022 Aug 24. PMID 36029884